CLINICAL TRIAL: NCT06165211
Title: The Effect of Nature-Based Sound Application on Fatigue and Patient Comfort in Hemodialysis Patients
Brief Title: Nature-Based Sound Application For Hemodialysis Patients
Acronym: NBSAFHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmiye ÇÖMLEKÇİ (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Necmiye ÇÖMLEKÇİ, Principal Investigator, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bartın Unıversity; 1919B012102111 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2023-05-30; First posted 2023-12-11 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Failure; Hemodialysis Patients; Fatigue; Patient Comfort; Nature Sounds
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature Sound Group (Experimental): During hemodialysis, 30 minutes with an Mp3 player and headphones (to minimize the effect of surrounding noise). Nature sounds consisting of bird, wind and tree sounds will be played.
  Interventions: Other: Nature sound listening
- Routine Care (Placebo Comparator): Patients will watch the program they want on the bedside TV during hemodialysis.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Nature sound listening — The intervention group listened to nature sounds for 30 minutes during hemodialysis. Nature sounds consisting of bird, wind and tree sounds will be played.
  Arms: Nature Sound Group
Other: Routine care — Patients will watch the program they want on the bedside TV during hemodialysis.
  Arms: Routine Care

SUMMARY:
Chronic renal failure is one of the most common chronic diseases in the world and in our country. Hemodialysis is the most commonly used treatment method in the treatment of chronic renal failure. In addition to its important benefits, hemodialysis treatment causes many problems such as fatigue, bone and joint pain, insomnia, mood disorders, sexual problems, paresthesia and nausea. In addition, patient comfort is adversely affected due to physical, psychosocial and environmental problems in hemodialysis patients. Elimination of symptoms in hemodialysis patients and ensuring patient comfort are important components of quality nursing care. For this purpose, it is reported that non-pharmacological evidence-based approaches such as listening to music, yoga, and exercise are used in the literature. Although there are studies examining the effectiveness of listening to music, the number of studies examining the effectiveness of nature-based sounds in hemodialysis patients is quite limited. It is known that sounds such as bird, ocean, water, wind sound have beneficial effects on human health in terms of physiological and psychosocial aspects. This project is to determine the effect of listening to nature sounds during hemodialysis treatment on fatigue and patient comfort.

Type of Study: The project was planned as a randomized controlled experimental study.

Population and Sample: The population of the study consists of patients who are treated in the Hemodialysis Unit of Bartin State Hospital. The sample was taken as d=0.80 power=0.90, α=0.05 and β=0.20, taking into account the data obtained from a similar study, and it was calculated as 30 patients in the intervention group and 30 patients in the control group, in total 60 patients.

Inclusion criteria for the study:

* To be receiving hemodialysis treatment for at least 6 months,
* Being over 18 years old,
* Not having a hearing and speaking disability,
* Not have a cognitive disability.

Exclusion criteria from the study:

* Receiving hemodialysis treatment for less than 6 months,
* Do not listen to the nature-based audio application for 30 minutes
* Being under the age of 18,
* Hearing and speech impairment,
* Having a cognitive disability.

DETAILED DESCRIPTION:
Data Collection Tools: Data will be collected using the Descriptive Information Form, Piper Fatigue Scale and Hemodialysis Patients Comfort Scale.

Descriptive Information Form: In this form, there are 15 questions created in line with the literature. It consists of two sections containing socio-demographic characteristics and disease information.

Piper Fatigue Scale (PFA): Piper et al. It was developed by in 1998. The scale consists of a total of 4 sub-dimensions and 22 items: behavioral sub-dimension (6 items), affective sub-dimension (5 items), emotional sub-dimension (5 items) and cognitive sub-dimension (6 items). Subscale scores and total fatigue scores are calculated using these 22 items. The other 5 items are used to calculate the subscales or total fatigue score. There are three open-ended questions to indicate the cause of fatigue. To calculate the score of the scale, the average score obtained from the scale is calculated by adding up all the scores of the 22 items and dividing by the number of items.

Hemodialysis Comfort Scale (HDCS): Hemodialysis Comfort Scale Orak et al. It was developed to determine the comfort levels of hemodialysis patients. The scale consists of a total of 9 items and two subscales: relaxation and coping. The total score evaluation of the scale and its sub-dimensions is determined by calculating the average score. Cronbach's alpha value of the scale was found to be 0.87.

Data Collection Process: The researcher will collect data in Bartin State Hospital Hemodialysis Unit and fill out the surveys using the interview method. while the patients are during the dialysis session in an average of 30-45 minutes. After the patients registered to the dialysis center are randomized by block randomization method as intervention and control groups, the Patient Diagnosis Form and pre-test (Piper Fatigue Scale and Hemodialysis Comfort Scale) will be applied to the patients before the hemodialysis session. Afterwards, during hemodialysis, listen with an Mp3 player and headphones (to minimize the effect of surrounding noise) for 30 minutes. Nature sounds will be played. After the hemodialysis session is completed, the patients will be given a posttest (Piper Fatigue Scale and Hemodialysis Comfort Scale) by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* To be receiving hemodialysis treatment for at least 6 months,
* Being over 18 years old,
* Not having a hearing and speaking disability,
* Not have a cognitive disability.

Exclusion Criteria:

* Receiving hemodialysis treatment for less than 6 months,
* Being under the age of 18,
* Hearing and speech impairment,
* Having a cognitive disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Piper Fatigue Scale Score | pre-intervention
  The scale consists of a total of 4 sub-dimensions and 22 items, including the behavioral sub-dimension (6 items), the affective sub-dimension (5 items), the sensory sub-dimension (5 items), and the cognitive sub-dimension (6 items). Subscale scores and total fatigue scores are calculated using these 22 items. The other 5 items are used to calculate the subscales or the total fatigue score. There are three open-ended questions to indicate the reason for fatigue. In order to calculate the score of the scale, the average score obtained from the scale is calculated by adding all the scores of 22 items and dividing them by the number of items.
Hemodialysis Comfort Scale Score | pre-intervention
  The scale consists of a total of 9 items and two sub-dimensions: relaxation and overcoming. The total score evaluation of the scale and its sub-dimensions is determined by calculating the average score.

SECONDARY OUTCOMES:
Piper Fatigue Scale Score | immediately after the intervention
  The scale consists of a total of 4 sub-dimensions and 22 items, including the behavioral sub-dimension (6 items), the affective sub-dimension (5 items), the sensory sub-dimension (5 items), and the cognitive sub-dimension (6 items). Subscale scores and total fatigue scores are calculated using these 22 items. The other 5 items are used to calculate the subscales or the total fatigue score. There are three open-ended questions to indicate the reason for fatigue. In order to calculate the score of the scale, the average score obtained from the scale is calculated by adding all the scores of 22 items and dividing them by the number of items.
Hemodialysis Comfort Scale Score | immediately after the intervention
  The scale consists of a total of 9 items and two sub-dimensions: relaxation and overcoming. The total score evaluation of the scale and its sub-dimensions is determined by calculating the average score.

CONTACTS AND LOCATIONS:
Overall Officials: Necmiye ÇÖMLEKÇİ, Principal Investigator — Bartın Unıversity
Locations (1):
- Necmiye ÇÖMLEKÇİ, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Research findings will be published with the article. In addition, research data, excluding personal data, will be shared for secondary results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared immediately after the research article is published.
Access Criteria: Data will be shared for secondary analyzes and meta-analysis studies.